CLINICAL TRIAL: NCT05418322
Title: The Effects of Oral Hygiene Interventions Prior Orthodontic Treatment in Adults-A Randomized Clinical Trial
Brief Title: The Effects of Oral Hygiene Interventions Prior Orthodontic Treatment in Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr. Lee Phey Ling, Principal investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PheyLing UMalaya
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Oral Hygiene; Adult
Keywords: Oral hygiene interventions; Adult; Prior orthodontic treatment

STUDY DESIGN:
Masking Description: The interventions and collection of data will be conducted by the same clinician. Therefore, both clinician and participants will not be blinded in this study given the nature of the interventions. However, as the participants will be randomized and allocated by an independent individual, blinding the clinician to the allocated interventions at the beginning of the trial, during baseline assessment, is possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal Oral Hygiene Intervention (Other): Each participant will be given oral hygiene instruction verbally by a clinician face to face.
  Interventions: Behavioral: Oral Hygiene Intervention
- Video-assisted Oral Hygiene Intervention (Other): Each participant will be required to watch a pre-recorded oral hygiene instruction video via a tablet in a separate room away from the clinician
  Interventions: Behavioral: Oral Hygiene Intervention

INTERVENTIONS:
Behavioral: Oral Hygiene Intervention — The oral hygiene instructions given in the two methods will be prepared in Bahasa Malaysia and English versions with the same content to avoid bias. The oral hygiene education will be validated by three dental specialists. A similar large dental teeth model and toothbrush will be used for the purpose of oral hygiene demonstration.

SUMMARY:
Orthodontic treatment has many recognized benefits such as enhancing esthetics and improving self-esteem in patients. However, like any other dental treatments, a successful orthodontic treatment requires patient cooperation, especially oral hygiene compliance.

Dental plaque that builds upon the orthodontic brackets in a poor oral environment consists of pathogenic biofilms that can lead to undesirable complications such as white spot lesions, gingivitis, and periodontal breakdown. Poor oral hygiene during orthodontic treatment often results in poor treatment quality and prolonged treatment duration. Fixed appliances increase the retention areas for plaque accumulation and this often makes maintaining good oral hygiene a challenge for the patients. Therefore, effective oral hygiene interventions are key in improving patients' knowledge, influencing good oral hygiene behaviors and ensuring patients can exercise good practices daily at home.

Oral hygiene education given to prospective orthodontic patients will allow them to understand their role and responsibilities in maintaining good oral care during treatment. This will help instill lasting good oral hygiene habits that can be maintained during the fixed appliance stage of treatment, thus reducing possible future treatment complications.

In this study, the investigators evaluate the effects of verbal and video-assisted oral hygiene interventions on patients' oral hygiene prior to orthodontic treatment.

DETAILED DESCRIPTION:
The present study evaluates the effectiveness of different oral hygiene interventions on patients' oral hygiene prior to orthodontic treatment.

Participants will be recruited from the Department of Pediatric Dentistry and Orthodontics, Faculty of Dentistry, University Malaya and will be selected from the postgraduate orthodontic treatment waiting list.

Patients meeting the selection criteria will be offered the opportunity to participate in the study during the visit prior to the orthodontic appliance placement. The participants will be equally distributed into two groups as follows:

Group 1: Verbal oral hygiene intervention

Group 2: Video-assisted oral hygiene intervention

A block randomization technique with 1:1 ratio of 5:5:5:5 fixed block sizes with no stratification will be used to randomly allocate the participants into the two interventions.

After baseline recording, full mouth supragingival scaling and treatments to remove any plaque retentive factor will be given to participants with the following measure:

i) Baseline full mouth plaque score >10% or ii) Baseline full mouth bleeding score >10%

Following treatment, each participant from group 1 will be given oral hygiene instruction verbally by a clinician face to face. In contrast, each participant from group 2 will be required to watch a pre-recorded oral hygiene instruction video via a tablet in a separate room away from the clinician. The oral hygiene instructions given in the two methods will be prepared in Bahasa Malaysia and English versions with the same content to avoid bias.

The aim of the study is to evaluate the effects of verbal and video-assisted oral hygiene interventions on patients' oral hygiene prior to orthodontic treatment.

The objectives of the study are:

1. To determine the changes in Full-mouth Plaque Score (FMPS) and Full-mouth Bleeding Score (FMBS) for both verbal and video groups after receiving oral hygiene instruction.
2. To compare the outcomes of Full-mouth Plaque Score (FMPS) and Full-mouth Bleeding Score (FMBS) between patients receiving verbal and video-assisted oral hygiene instruction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Plan to undergo orthodontic treatment and is eligible for orthodontic treatment with fixed appliances.
* Clinical gingival health (<10% bleeding score) or localized gingivitis (10%-30% bleeding score) or generalized gingivitis (>30% bleeding score)
* Presence of BPE code 0/1/2 with no obvious evidence of interdental recession
* Have at least 20 teeth
* Able to understand Bahasa Malaysia and English languages

Exclusion Criteria:

* Presence of BPE code 3/4
* Current or previous history of periodontitis
* Smokers
* Severe or chronic illnesses (such as diabetes, cardiovascular diseases, stroke, etc)
* Physically impaired
* Orofacial deformities
* History of previous orthodontic treatment
* Intake of antibiotics within 6 months before and during the study period
* Taking drugs that influence gingival inflammation or bleeding (eg anticoagulants, cortisone)
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Changes between the Full Mouth Plaque Score(FMPS) measurement at baseline (T0), at 2 weeks (T1), and at 4 weeks (T2) after the intervention | Baseline, 2 weeks and 4 weeks
  Presence or absence of plaque deposits on each tooth surface (mesial, distal, buccal and lingual/palatal) in the dentition is recorded in a dichotomous manner. The plaque deposits will be disclosed using a disclosing solution to facilitate their detection. The presence of plaque is recorded in a plaque chart.

SECONDARY OUTCOMES:
Changes in Full Mouth Bleeding Score (FMBS) at baseline (T0) and at 4 weeks post intervention (T2) | Baseline and 4 weeks
  Presence or absence of gingival bleeding on each tooth surface (mesial, distal, buccal and lingual/palatal) in the dentition is recorded in a dichotomous manner. The FMBS will be performed through gentle probing of the gingival crevice on each tooth surface. A positive finding will be recorded if bleeding occurs within 10 seconds. The presence of bleeding is recorded in a FMBS chart.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Malaya, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Lew KK. Attitudes and perceptions of adults towards orthodontic treatment in an Asian community. Community Dent Oral Epidemiol. 1993 Feb;21(1):31-5. doi: 10.1111/j.1600-0528.1993.tb00715.x. PMID 8432102
- [Background] Axelsson P, Nystrom B, Lindhe J. The long-term effect of a plaque control program on tooth mortality, caries and periodontal disease in adults. Results after 30 years of maintenance. J Clin Periodontol. 2004 Sep;31(9):749-57. doi: 10.1111/j.1600-051X.2004.00563.x. PMID 15312097
- [Background] Soldo M, Matijevic J, Malcic Ivanisevic A, Cukovic-Bagic I, Marks L, Nikolov Boric D, Jukic Krmek S. Impact of oral hygiene instructions on plaque index in adolescents. Cent Eur J Public Health. 2020 Jun;28(2):103-107. doi: 10.21101/cejph.a5066. PMID 32592553
- [Background] Cardoso Mde A, Saraiva PP, Maltagliati LA, Rhoden FK, Costa CC, Normando D, Capelozza Filho L. Alterations in plaque accumulation and gingival inflammation promoted by treatment with self-ligating and conventional orthodontic brackets. Dental Press J Orthod. 2015 Mar-Apr;20(2):35-41. doi: 10.1590/2176-9451.20.2.035-041.oar. PMID 25992985